CLINICAL TRIAL: NCT02756377
Title: A Comparison of Mouth Rinse Containing Alcohol-free Chlorhexidine With a Cetylpyridinium Chloride in Periodontal Diseases (A Randomized, Double-blind Clinical Trials)
Brief Title: A Comparison of Mouth Rinse Containing Alcohol-free Chlorhexidine With a Cetylpyridinium Chloride in Periodontal Diseases
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Islamic Azad University, Sanandaj (Other)
Responsible Party: Principal Investigator, Amirhossein Farahmand, clinical effectiveness of 0.05% cetylpyridinium chloride mouth rinse in patients with gingivitis as compared to non-alcoholic chlorhexidine mouth wash, Islamic Azad University, Sanandaj
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 483
Record Dates: First submitted 2016-04-27; First posted 2016-04-29 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cetylpyridinium chloride (Active Comparator): mouthwash (cetylpyridinium chloride)10 ml by patients routinely washed two times in one day for about 30 seconds for two weeks.
  Interventions: Drug: cetylpyridinium chloride mouthwash; Drug: Chlorhexidine mouthwash
- Chlorhexidine mouthwash (Active Comparator): mouthwash ( Alcohol-free chlorhexidine)10 ml by patients routinely washed two times in one day for about 30 seconds for two weeks.
  Interventions: Drug: cetylpyridinium chloride mouthwash

INTERVENTIONS:
Drug: cetylpyridinium chloride mouthwash — cetylpyridinium chloride mouthwash, 10 ml by patients routinely washed two times in one day for about 30 seconds for two weeks.
  Other Names: control
Drug: Chlorhexidine mouthwash — Chlorhexidine mouthwash,10 ml by patients routinely washed two times in one day for about 30 seconds for two weeks.
  Other Names: Experimental Chlorhexidine mouthwash made by Perio-Kin, Livar CO. Spain
  Arms: cetylpyridinium chloride

SUMMARY:
Aim: clinical effectiveness of 0.05% cetylpyridinium chloride mouth rinse in patients with gingivitis as compared to non-alcoholic chlorhexidine mouth wash.

Methods & Material: Twenty-four subjects, without systemic diseases, with plaque-induced gingivitis will be selected for this study. The patients were treated with scaling and root planing at the baseline; Oral hygiene instructions were given that included brushing twice- daily, The volunteers brushed their teeth with the Bass brushing technique for at least 2 minutes, these patients were randomly ,equally divided into two groups, Group A: perform daily mouthwashes twice a day with the solution containing 10 ml of 0.05 cetyl pyridinium, (Vi-one, Rojin, Cosmetic-Lab, Kurdistan -Iran), Group B: use daily mouthwashes twice a day with 10ml of the chlorhexidine(Kin Laboratories, Spain), On day 0,7,15 and day 21 of each phase the Plaque Index (PI), Pocket depth(PD), Stain Index(SI) and Bleeding Index (BI) of each volunteer were measured.

DETAILED DESCRIPTION:
In this study, 34 patients referred to periodontics Department that no serious systemic disease in terms of periodontitis and disease Gingivitis (ie pockets of periodontal tissue to a depth of less than or equal to 4 mm without CAL in the jaw down or up) the following explanation necessary for the procedure tastings consent, the index of oral hygiene (plaque index) index # Turesky, pocket depth and to control the inflammatory condition * bleeding index bleeding during the probe based on Carter and Barnes (if any bleeding number 1 and its absence 0) and attachment loss were evaluated areas. The amount of pigment (Stain) after of using mouthwash based on S.I (Stain Index) was evaluated .

ELIGIBILITY:
Inclusion Criteria:Inclusion criteria: adult patients with gingivitis, older than 18 years old, systemically healthy, and having at least 20 teeth.

Exclusion Criteria:patients with cavitated caries, no periodontal pockets larger than 4 mm, orthodontic appliances or removable prostheses, allergies to cetyl pyridinium or CHX, use of antibiotics and anti-inflammatory drugs in the past 3 months that might alter normal gingival health, oral prophylaxis outside of study; use of oral chlorhexidine products or participation in an oral rinse study within 3 months prior to baseline examination, pregnancy or nursing, smoking.

Study Population 34 eligibles were enrolled in the study, was designed as a Randomized, Double-blind clinical trials.

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2014-05; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Reduction of bleeding on probing | 7 days
  Periodontal pobe

SECONDARY OUTCOMES:
Reduction of plaque index | 7 days
  Plaque Index (O'Leary)
Reduction of pocket depth | 7days
  Periodontal pobe

IPD SHARING:
Plan to Share IPD: No